CLINICAL TRIAL: NCT02830373
Title: Chinese Registry of Assisted Embolization for Unruptured Wide Necked Intracranial Aneurysm Using LVIS Stent
Acronym: CRANIAL-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Qinghai Huang, Deputy Director of Neurosurgery, Clinical Professor, Changhai Hospital
Other Study IDs: CHEC2016-058
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Self Efficacy; Medical Device Complication
Keywords: LVIS stents; Intracranial aneurysm; Unruptured aneurysm; Wide-necked aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LVIS stents group: patients with unruptured intracranial saccular aneurysms which located in the internal carotid artery or vertebra-basilar artery will be treated with a LVIS stent with coils
  Interventions: Device: LVIS stents

INTERVENTIONS:
Device: LVIS stents — Patients who meet the inclusion criteria will be treated with a low profile visualized intraluminal support (LVIS) stent with coils.

SUMMARY:
This study aims to investigating the efficacy and safety of low profile visualized intraluminal support (LVIS) stents for the treatment of unruptured intracranial saccular aneurysms.

DETAILED DESCRIPTION:
This study is a prospective multi-centre observational single-arm clinical trial, aiming to investigating the efficacy and safety of low profile visualized intraluminal support (LVIS) stents combined with coils for the treatment of unruptured intracranial saccular aneurysms. As the protocol, clinical follow-up at 30 days (±7 days) after procedure, DSA or MRA follow-up at 6 months (±30 days) after procedure, and clinical follow-up at 1 year (±30 days) after procedure was conducted for each patient. The primary end-points include major adverse events (cerebral infarct and death) in 30 days post-procedure, complete occlusion rate at 6 months (180±30d) follow-up. The secondary end-points were immediate technical success (successful device placement) rate, immediate complete occlusion rate, recurrence rate at 6 months (180±30d) follow-up and in-stent stenosis or obliteration rate at 6 months (180±30d) follow-up. Duration of this study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all the following criteria will be enrolled:

  1. Patients of the age 18-75 years old.
  2. Patients diagnosed with unruptured intracranial saccular aneurysms via CTA, MRA or DSA.
  3. Patients treated with LVIS stents combined with coils.
  4. Patients willing to follow the clinical trial instructions and receive follow-up assessment.
  5. Patients accepting to participate to the study and sign the consent forms.

Exclusion Criteria:

* Patients meeting any following criterion will be excluded:

  1. Patients without proper artery approach.
  2. Patients with AVM.
  3. Patients with a fusiform or dissecting aneurysm.
  4. Patients with a recurrent aneurysm.
  5. Patients treated with a LVIS stent without coils.
  6. Patients in poor clinical status, with mRS ≥4.
  7. Patients with life expectancy less than 12 months.
  8. Patients participated in other clinical trial, while has not reach the primary endpoint.
  9. Patients can not accept anti-platelet regimen.
  10. Patients allergic to contrast agent or intolerable.
  11. Patients whom the researchers consider should not participate in or continue this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population was the patients with unruptured intracranial saccular aneurysms which located in the internal carotid artery or vertebra-basilar artery.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse events (cerebral infarct, death) in 30 days post the procedure | During 30 days post the procedure
  Major adverse events (cerebral infarct, death) in 30 days post the procedure is defined as post-procedural cerebral infarct or death caused by any reasons
Complete occlusion rate at 6 months (180±30d) follow-up | At 6 months (180±30d) follow-up
  Complete occlusion at 6 months follow-up is defined as 100% occlusion of aneurysmal sac proved by DSA at 6 months follow-up

SECONDARY OUTCOMES:
Immediate technical success rate (successful device placement) | Within 24 hours postoperatively
  Immediate technical successful is defined as good apposition of stents, effective coverage of aneurysmal neck proved by post-procedural imaging examination.
Immediate complete occlusion rate | Within 24 hours postoperatively
  Immediate Raymond scale is defined as immediate angiographic result according to the simplified Raymond scale, classⅠ: complete occlusion; class Ⅱ: neck remnant; class Ⅲ: incomplete occlusion.
Recurrence rate at 6 months (180±30d) follow-up | At 6 months (180±30d) follow-up
  Recurrence rate: defined as increased contrast filling into the aneurysmal sac compared with immediate angiographic result.
In-stent stenosis or obliteration rate at 6 months (180±30d) follow-up | At 6 months (180±30d) follow-up
  In-stent stenosis at 6 months follow-up is defined as stenosis more than 50% proved by DSA at 6 months follow-up. In-stent occlusion or thrombosis at 6 months follow-up is defined as complete occlusion of the stent proved by DSA at 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Doctor, Principal Investigator — Department of Neurosurgery, Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong Y, Wang YJ, Deng Z, Wu Q, Zhang JM. Stent-assisted coiling versus coiling in treatment of intracranial aneurysm: a systematic review and meta-analysis. PLoS One. 2014 Jan 15;9(1):e82311. doi: 10.1371/journal.pone.0082311. eCollection 2014. PMID 24454690
- [Background] Geyik S, Yavuz K, Yurttutan N, Saatci I, Cekirge HS. Stent-assisted coiling in endovascular treatment of 500 consecutive cerebral aneurysms with long-term follow-up. AJNR Am J Neuroradiol. 2013 Nov-Dec;34(11):2157-62. doi: 10.3174/ajnr.A3574. Epub 2013 Jul 25. PMID 23886748
- [Background] Poncyljusz W, Bilinski P, Safranow K, Baron J, Zbroszczyk M, Jaworski M, Bereza S, Burke TH. The LVIS/LVIS Jr. stents in the treatment of wide-neck intracranial aneurysms: multicentre registry. J Neurointerv Surg. 2015 Jul;7(7):524-9. doi: 10.1136/neurintsurg-2014-011229. Epub 2014 May 14. PMID 24827067
- [Result] Feng Z, Fang Y, Xu Y, Hong B, Zhao W, Liu J, Huang Q. The safety and efficacy of low profile visualized intraluminal support (LVIS) stents in assisting coil embolization of intracranial saccular aneurysms: a single center experience. J Neurointerv Surg. 2016 Nov;8(11):1192-1196. doi: 10.1136/neurintsurg-2015-012090. Epub 2016 Jan 8. PMID 26747876
- [Result] Fiorella D, Arthur A, Boulos A, Diaz O, Jabbour P, Pride L, Turk AS, Woo HH, Derdeyn C, Millar J, Clifton A. Final results of the US humanitarian device exemption study of the low-profile visualized intraluminal support (LVIS) device. J Neurointerv Surg. 2016 Sep;8(9):894-7. doi: 10.1136/neurintsurg-2015-011937. Epub 2015 Sep 21. PMID 26391016
- [Result] Cho YD, Sohn CH, Kang HS, Kim JE, Cho WS, Hwang G, Kwon OK, Ko MS, Park NM, Han MH. Coil embolization of intracranial saccular aneurysms using the Low-profile Visualized Intraluminal Support (LVIS) device. Neuroradiology. 2014 Jul;56(7):543-51. doi: 10.1007/s00234-014-1363-x. Epub 2014 Apr 17. PMID 24740581